CLINICAL TRIAL: NCT07227766
Title: Dietary Reversal of the Reprometabolic Syndrome
Acronym: LFD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-1702
Record Dates: First submitted 2025-11-11; First posted 2025-11-13 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Obesity & Overweight; Infertility, Female
Keywords: Infertility; Reproductive Hormones; Low-Fat Diet; Obesity; Hypothalamic-pitutary-ovarian axis
MeSH Terms: conditions — Obesity; Overweight; Infertility, Female; Infertility | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-Fat Diet (Experimental): Participants will eat a customized, eucaloric low-fat diet for one month
  Interventions: Dietary Supplement: Low-fat diet

INTERVENTIONS:
Dietary Supplement: Low-fat diet — Participants will eat a one-month eucaloric high-fat diet.

SUMMARY:
This study proposes to test the specific question that a eucaloric, low-fat diet given to women with obesity will result in an increase in reproductive hormones.

DETAILED DESCRIPTION:
This an open-label, multi site study in pre-menopausal women aged 18-40 years old with a history of regular menstrual cycles (25-35 days long) of high BMI. The objective of the study will be to determine the effects of a one month long, eucaloric low-fat diet on reproductive hormone levels in women with a high BMI. The study will occur over 4 menstrual cycle (approximately 4 months). During the study the participants will have a pre-diet cycle where no food will be consumed, an on-diet cycle where the customized low-fat diet will be consumed, and two post diet cycles. First morning voided urine will be collected during all four cycles along with 3 blood draws during the study. Participants will be asked to use a reliable barrier method of birth control or abstain from intercourse during the study.

ELIGIBILITY:
Inclusion Criteria:

* Normal TSH and prolactin
* Regular menstrual cycles every 25-40 days
* No history of chronic disease affecting hormone production, metabolism or clearance
* No use of reproductive hormones, or medications/supplements known to impact them, within 3 months of enrollment
* Use of a reliable method of contraception (female or male partner sterilization, IUD, abstinence, diaphragm or cervical cap)
* Normal ovarian reserve (AMH of 0.5ng/ml or greater)
* Normal testosterone levels at screening or absence of clinical evidence of hyperandrogenemia (acne, facial hirsutism [defined as Ferriman-Gallwey score>8] or alopecia)

Exclusion Criteria:

* Baseline dietary assessment indicative of 28% or less daily calories from fat
* Inability to comply with the protocol (many meals per week eaten outside of the home, frequent travel)
* Pregnancy or planned pregnancy within next 6 months at time of screening
* HbA1C >6.5%

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study examines female reproductive hormones.
Enrollment: 30 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Urinary Pregnadiol Glucouronide concentration in ug/mg creatinine | From enrollment for 4 months post enrollment

SECONDARY OUTCOMES:
Amount of Urinary estrogen | From enrollment to 4 months
  Urinary estrogen concentration in microgram/mg of Creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Nanette Santoro, MD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided